CLINICAL TRIAL: NCT03115242
Title: Contrast Enhanced Ultrasound of Carotid Plaque in Acute Ischemic Stroke
Acronym: CUSCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: Jennifer YEUNG (neurologist) (Unknown); Aurélien MAURIZOT (angiologist) (Unknown); Simon CHABAY (angiologist) (Unknown); Daniela STANCIU (neurologist) (Unknown)
Responsible Party: Principal Investigator, Dr Jean-Michel BAUD, Investigator coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P14/06_CUSCAS; 2014-A01181-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-09-05; First posted 2017-04-14 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute ischemic carotid stroke (Experimental): Patients hospitalized in the neurovascular intensive care unit for an acute ischemic stroke with a carotid plaque responding to inclusion criteria.
  These patients receive a contrast injection Sonovue® will be performed during the neck vessels doppler ultrasound.
  Interventions: Other: Contrast injection Sonovue®

INTERVENTIONS:
Other: Contrast injection Sonovue® — In addition to standardized assessment routine care, a contrast injection will be performed during the neck vessels doppler ultrasound.

SUMMARY:
This is a biomedical, single-center, and prospective study of a consecutive patients cohort in acute ischemic stroke with carotid plaque.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the prevalence of the contrast taking carotid plaques in these acute ischemic strokes.

The secondary objectives are:

* to determine the clinical, sonographic, CT scanner and MRI characteristics of patients in constituted acute cerebral ischemia with carotid atherosclerotic plaque taking contrast to the doppler ultrasound.
* to explore of the plaque contrast enhancement at 6 months (new injection).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged at least 18 years hospitalized with ischemic stroke signs in the carotid territory, objectified on brain MRI with positive DWI.
* Carotid plaque > 2.5 mm thickness in the ipsilateral carotid territory to the AIC, low echogenicity (Type 1, 2, 3, and 4a of the classification Geroulakos) measured by the assessment "GSM" (median gray level).
* Free and informed consent patient or his representative for contrast injection microbubble.
* Affiliated to health insurance.

Exclusion Criteria:

* Severe cerebral infarction with NIHSS> 25
* No-indications to the contrast medium injection
* Recent myocardial infarction, unstable angina.
* Heart failure stage III / IV New York Heart Association.
* Cardiac shunt left-right, respiratory distress.
* Allergy to albumin or contrast agents.
* Carotid plaques and hyperechoic calcified (however these plaques will be counted to determine their prevalence in acute AIC).
* Carotid dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement of carotid plaque prevalence in ultrasound doppler | Day 1

SECONDARY OUTCOMES:
Patient's demographics data | Day 1
Patient's sonographic and MRI characteristics. | Day1
  confirmation of the recent character of stroke on the DWI, search for stroke sequelae and white matter disease on the FLAIR, search of the thrombus on the T2*, search occluded artery on the 3DTOF
describe the aspect of the carotid plaque on CT angiography. | between 1 to 5 days
  NASCET stenosis and the aspect (smooth, irregular, ulcerated)
Persistence , decrease or loss of contrast enhancement in ultrasound doppler. | Month 6
Cerebral infarction recurrence | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer YEUNG, Neurologist, Principal Investigator — Versailles Hospital; Jean-Michel BAUD, Angiologist, Principal Investigator — Versailles Hospital; Aurélien MAURIZOT, Angiologist — Versailles Hospital; Simon CHABAY, Angiologist — Versailles Hospital; Daniela STANCIU, Neurologist — Versailles Hospital
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Undecided